CLINICAL TRIAL: NCT06609473
Title: Proof-of-Concept Testing of the Cardiovascular Health Equity Through Food (CHEF) Intervention in Childhood Cancer Survivors
Acronym: CHEF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Rahela Aziz-Bose, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 24-423
Record Dates: First submitted 2024-09-20; First posted 2024-09-24 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Childhood Cancer; Childhood Cancer Survivors
Keywords: Cardiovascular Health; Childhood Cancer; Childhood Cancer Survivorship
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CHEF Program (Experimental): Enrolled participants and caregivers will complete:
  * Baseline visit and survey
  * Meeting with a certified benefits counselor by phone or video teleconference
  * Kitchen equipment delivery
  * Weekly meal kit deliveries
  * Monthly grocery support via gift card
  * Second meeting with a certified benefits counselor
  * 3-month survey
  * Final survey and interview with study staff
  Interventions: Behavioral: CHEF Intervention Program

INTERVENTIONS:
Behavioral: CHEF Intervention Program — Poverty-targeted intervention utilizing direct resource provision of healthy meal kits and groceries, as well as assisted referral and enrollment in government nutrition assistance benefits, SNAP (Supplement Nutrition Assistance Program) and/or WIC (Woman, Infants, and Children Program). Meal kits will be delivered by a commercial meal kit vendor. Grocery gift cards will be delivered via email, mail, or in-person. Kitchen equipment will be delivered to caregiver residence.
  Other Names: Cardiovascular Health Equity Through Food Program

SUMMARY:
The goal of the Cardiovascular Health Equity Through Food (CHEF) program is to make it easier for participants and families to cook and eat healthy foods during and following childhood cancer treatment with the long-term goal of supporting heart health.

DETAILED DESCRIPTION:
This is a proof-of-concept study to test the CHEF intervention by utilizing survey, interview, and medical record data from participants with cancer to determine the intervention's impact on cardiovascular-relevant outcomes and to identify optimal implementation strategies for the intervention.

The research study procedures include screening for eligibility, questionnaires, and a brief interview.

Participation in this research study is expected to last 6 months.

It is expected about 17 participants/families will participate in this research study.

ELIGIBILITY:
Inclusion Criteria:

* Child with any primary cancer diagnosis (non-relapsed, non-secondary malignancy) who has received cancer-directed therapy that includes chemotherapy and/or radiation therapy;
* Child is within one of the following time windows:

  1. Among those receiving chemotherapy, any time from start of last planned cycle of chemotherapy until 12 months from completion of chemotherapy;
  2. Among those receiving radiation therapy alone or radiation and surgery, any time from completion of radiation until 12 months post completion;
* Child has 1 or more cardiovascular risk factor (defined as any of: body mass index ≥ 85th percentile; systolic or diastolic blood pressure ≥90th percentile; dyslipidemia [triglycerides ≥150 mg/dL, total cholesterol ≥200 mg/dL, LDL cholesterol ≥130 mg/dL, HDL cholesterol ≤40 mg/dL]; impaired glucose metabolism [fasting glucose ≥100 mg/dL, hemoglobin A1c ≥5.7%]; anthracycline exposure ≥100 mg/m2; or any radiation exposure to chest, brain, thoracic spine, or total body);
* Child is ≤18 years of age at time of enrollment, or over 18 years of age but under medical guardianship;
* Parent/guardian screened positive for food insecurity.* *Assessed through validated 2-item food insecurity screen.

Exclusion Criteria:

* Patient received only surgery, or watchful waiting/surveillance, for cancer- directed therapy;
* Foreign national family receiving cancer care as an embassy-pay patient.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 17 (Estimated)
Dates: Start 2025-04-07 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2028-02-28 (Estimated)

PRIMARY OUTCOMES:
Change in Dietary Quality Score | From baseline to 6 months
  The change in mean participant dietary quality from study period T1 (baseline) to study period T3 (month 6), as measured by the Rapid Prime Dietary Quality Score Screener (scored 0-52, higher score indicates higher quality diet).

SECONDARY OUTCOMES:
Change in Food Security Status | From baseline to 6 months
  Change in the proportion of participants reporting any food insecurity from study period T1 (baseline) to study period T3 (month 6), as measured by the Abbreviated Child and Adult Food Security Survey (ACAFSS).
Proportion of Providers Consenting to Participant Approach | Up to 9 months per enrollment period
  Defined as the number of providers consenting to participant/caregiver approach for study enrollment out of the number of providers contacted to request permission to approach. A positive response from the provider will be required for the study team to approach participant/caregivers.
Consent Rate | Up to 9 months per enrollment period
  Defined as the proportion of eligible participants/caregivers approached for consent who are enrolled in the study.
Retention | From baseline to 6 months
  Defined as the proportion of participants who remain enrolled in the study at each study timepoint from study period T1 (baseline) to study period T3 (6 months).
Utilization Rate of Benefits Assistance | Up to 6 months
  Defined as the number of participants/caregivers requesting assistance with SNAP (Supplemental Nutrition Assistance Program) and/or WIC (Women, Infants, and Children Program) benefits.
Intervention Fidelity | Up to 6 months
  Defined as proportion of meal kits delivered, proportion of meal kits prepared, proportion of meal kits consumed, and number of unplanned modifications of intervention delivery of meal kits, kitchen equipment, or gift cards.

OTHER OUTCOMES:
Change in Dietary Quality DietID Score | From baseline to 6 months
  The change in mean participant dietary quality from study period T1 (baseline) to study period T3 (month 6), as measured by DietID Healthy Eating Index 2020 score (scored 0-100, higher score indicates higher quality diet).
Change in Food Insecurity Severity | From baseline to 6 months
  Change in severity of participant/household food insecurity from study period T1 (baseline) to study period T3 (month 6) will be assessed using number of affirmative responses on the 8-item Abbreviated Child and Adult Food Security Survey; a higher number of affirmative responses indicates lower food security.

CONTACTS AND LOCATIONS:
Overall Officials: Rahela Aziz-Bose, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Boston Children's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: Rahela Aziz-Bose (PI) [rahela_aziz-bose@dfci.harvard.edu]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu